CLINICAL TRIAL: NCT05939115
Title: Efficacy of Unilateral Versus Bilateral Accelerated Theta Burst Stimulation in Treatment of Patients With Bipolar Depression and Suicidality
Brief Title: Intensive Accelerated Theta Burst Stimulation in Treatment of Patients With Bipolar Depression and Suicidality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Medhat Bassiony, Professor of Psychiatry, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9697
Record Dates: First submitted 2023-06-24; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Left unilateral aTBS (Active Comparator): Participants who are randomly assigned to this group will receive iTBS (intermittent theta burst stimulation) to the left dorsolateral prefrontal cortex (LDLPFC) determined using Beam method for 1800 pulses with an intertreatment interval of fifty minutes. Stimulation was at 90% of resting motor threshold. Patients received ten sessions every day for five consecutive days for a total of fifty sessions (90,000 pulses).
  Interventions: Device: Transcranial Magnetic Stimulation MagPro R30 with the MCF-B70 figure-of-eight coil (MagVenture, Denmark)
- Sequential bilateral aTBS (Active Comparator): Participants who are randomly assigned to this group will receive ten sessions daily for five consecutive days for a total of fifty sessions. During each session continuous theta burst stimulation (cTBS) in which (1800 pulses) are delivered continuously over 120 seconds to the right dorsolateral prefrontal cortex (RDLPFC) is administered first, followed by iTBS in which 1800 pulses are delivered in 2 second bursts, repeated every 10 seconds for 570 seconds (1800 pulses) to the left dorsolateral prefrontal cortex (LDLPFC) with using beam method for target localization. Stimulation was at 90% of resting motor threshold.
  Interventions: Device: Transcranial Magnetic Stimulation MagPro R30 with the MCF-B70 figure-of-eight coil (MagVenture, Denmark)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation MagPro R30 with the MCF-B70 figure-of-eight coil (MagVenture, Denmark) — TMS Therapy System with Theta Burst Stimulation

SUMMARY:
The objective of this study is to compare the efficacy of left unilateral versus bilateral accelerated Theta Burst Stimulation (TBS) in suicidal reduction and in reduction of severity of depressive symptoms in patients with bipolar depression.

DETAILED DESCRIPTION:
Introduction:

Repetitive transcranial magnetic stimulation (rTMS) therapy is a noninvasive neurostimulation treatment that has been adopted as a first-line treatment for pharmacotherapy-resistant major depressive disorder (MDD) (Milev et al., 2016). rTMS induces electrical activity in the cortex using magnetic fields generated outside of the head. However, the evidence for antidepressant efficacy of rTMS in the treatment of bipolar depression is limited and derived primarily from small trials (Tavares et al., 2017, Dolberg et al., 2002, Nahas et al., 2003, Beyne et al., 2014, Tamas et al., 2007) and subsets of trials in major depression that included individuals with bipolar disorder (McGirr et al., 2016, Nguyen et al., 2021 ).

The proposed study will examine sequential bilateral versus Unilateral accelerated theta burst stimulation (aTBS) in treatment of patients with bipolar depression and suicidality.

Hypothesis:

We assume that bilateral accelerated TBS is superior than left unilateral accelerated TBS in treatment of suicidality while bilateral accelerated TBS is as effective as left unilateral accelerated TBS in treatment of depressive symptoms in bipolar patients.

Aim:

This study aims to reduce morbidity and mortality of bipolar depressive patients and to improve overall functioning.

Objectives:

1. To compare efficacy of left unilateral versus bilateral accelerated TBS in suicidal reduction in patients with bipolar depression.
2. To compare efficacy of left unilateral versus bilateral accelerated TBS in reduction of severity of depressive symptoms in bipolar disorder as well as response and remission rates.
3. To investigate association between the reduction of suicidality and the reduction of depressive symptoms

Subjects and methods

1. Technical design:

   Site of the study: psychiatric department TMS Unit at Zagazig University Hospital

   Sample size:

   Assuming that Percent of improvment of depression scale in bipolar patients ( response rate) in unilateral TMS was 47% and bilateral TMS was 80% (Kazemi et al.,2016) so at power of study 80% and confidence interval 95%, the sample size was calculated to be 58 cases ( 29 in each group) ( Open Epi )
   * The samples will be allocated randomly into two groups (1:1) :
   * First group: will be treated by left unilateral accelerated TBS
   * Second group: will be treated by bilateral accelerated TBS
2. Operational design

   * Study design:
   * Open label randomized clinical trial with two parallel treatment arms
   * Methods:
   * Patients will be allocated randomly into two groups (1:1).
   * The randomization scheme was generated by using the Web site Randomization.com ⟨http://www.randomization.com⟩.
   * Group 1 will receive (left unilateral aTBS); group 2 will receive ( bilateral aTBS)
   * Device: MagPro R30 with the MCF-B70 figure-of-eight coil (MagVenture, Denmark)
   * Details of treatment sessions:
   * Group 1 (left unilateral aTBS): "Active comparator"
   * They will receive accelerated iTBS. Stimulation with F-8 coil was administered to the left dorsolateral prefrontal cortex (DL-PFC) determined using Beam method. Stimulation was at 90% MT intermittent theta burst (iTBS) for 1800 pulses with an intertreatment interval of fifty minutes. Patients received ten sessions every day for five consecutive days for a total of fifty sessions (90,000 pulses).
   * Group 2 ( bilateral aTBS) : "Active comparator"
   * Bilateral accelerated theta burst stimulation (aTBS). Ten sessions are administered daily for five consecutive days for a total of fifty sessions .During each session continuous theta burst stimulation (cTBS) in which (1800 pulses) are delivered continuously over 120 seconds to the right dorsolateral prefrontal cortex (RDLPFC) is administered first, followed by iTBS in which 1800 pulses are delivered in 2 second bursts, repeated every 10 seconds for 570 seconds (1800 pulses) to the left dorsolateral prefrontal cortex (LDLPFC) with using beam method for target localization .
   * The theta burst stimulation (TBS) parameters were adopted from prior work, with 3-pulse 50 Hz bursts given every 200 ms (at 5 Hz) with an intensity of 90% of resting motor threthold (RMT)
   * Motor threshold: Using single pulse TMS, the scalp position of lowest motor threshold over primary motor cortex to produce visual contraction of the first dorsal (thumb) interosseous or abductor pollicis brevis muscle . Resting motor threshold (MT) was defined using the Adaptive Pest online algorithm.

Participants :

All the participants who will be enrolled in the study will be subjected to the following:

1. A semi-structured interview will be employed to obtain socio-demographic and clinical data.
2. Psychometric tools:

The scales will be done at baseline and at the end of each day of five treatment days .

1. Montgomery-Asberg depression rating scale (MADRS)
2. The Beck Depression Inventory
3. Columbia Suicide Severity Rating Scale (C-SSRS)
4. Young Mania Rating Scale (YMRS)

Administrative design

* Approval was obtained from the Institutional Review Board (IRB) and the Department of Psychiatry, Zagazig University, Egypt.
* A written consent will be signed by the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major depressive episode as a part of bipolar (I or II) disorder and confirmed by Structured Clinical Interview for DSM-IV-TR Axis I Disorders (SCID-I)
* Meet the threshold on the total MADRS score of >/=35 at baseline visit (severe)
* Meet the threshold on the total BDI-II score of >/=30 at baseline visit (severe)
* Ongoing suicidal ideation and/or behavior (confirmed with Columbia Scale for the Rating of Suicide Severity (C-SSRS) , score >/=3 (moderate to high risk)
* Age 19 years or older (Adults, Older Adults)
* Right handedness
* Both genders
* Able to provide informed consent to participate in the study
* Participants were required to have been taking a stable pharmacological regimen for 2 weeks before screening that had to include a mood stabilizer (lithium >0.6 mEq/L or valproate >350 mM/L), an atypical antipsychotic, or a combination of a mood stabilizer and an atypical antipsychotic. For participants with BD type II, lamotrigine monotherapy was acceptable if the dose was greater than 100 mg daily
* Pass the TMS adult safety screening (TASS) questionnaire

Exclusion Criteria:

* No current substance abuse disorder for the past 3 months (previous substance abuse not exclusionary)
* Any psychotic disorder or current active psychotic symptoms
* No dementia or other major neurological disorders
* No major medical illness, for example metastatic cancer, end stage renal disease
* Not able to verify contact information. Participants must be able to follow through with the study & must have verified contact information and at least one verified contact
* Pregnancy. While there are no known risks to a fetus this is a new use of TMS, which has not been tested, thus pregnancy is exclusionary
* Any history of any clinically significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes
* Conductive, ferromagnetic or other magnetic sensitive metals that are implanted or are non-removable within 30 cm treatment coil (around the head)
* Score on Young Mania Rating Scale (YMRS) greater than 12 (patients with mixed features have been shown not to respond well to TMS treatment)
* Rapid cycling Bipolar illness (patients with > 4 mood episodes within the past year will be excluded, as they have a higher risk of switch to mania)
* Non response to ECT in current episode.
* Current severe insomnia (must sleep a minimum of 5 hours the night before stimulation)
* Are currently (or in the last 4 weeks) taking lorazepam greater than 2 mg daily (or equivalent) due to the potential to limit rTMS efficacy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal ideation and behaviors as measured by Columbia Suicide Severity Rating Scale (C-SSRS) | Assessed at baseline (day 0) , post-inpatient treatment completion (day 5) , 1 month ,3 month and 6 month.
  The SI severity scale is composed of five yes=no questions of increasingly severe suicidal thoughts: a wish to be dead (1), non-specific suicidal thoughts (2), suicidal thoughts with a method (3), suicidal intent without specific plan (4), and suicidal intent with specific plan (5).
  This scale was scored from 0 to 5 according to the most severe suicidal ideation endorsed. Higher scores mean worse outcome.
  Suicidal behaviors were assessed dichotomously (yes=no) and include actual suicide attempts, interrupted suicide attempts, aborted suicide attempts, other preparatory acts (e.g., collecting pills, writing suicide note), and non-suicidal self-injury (NSSI).

SECONDARY OUTCOMES:
Change from baseline Montgomery-Åsberg Depression Rating Scale (MADRS) Score | Assessed at baseline (day 0) , post-inpatient treatment completion (day 5) , 1 month ,3 month and 6 month.
  The Montgomery-Åsberg Depression Rating Scale (MADRS), is a ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  Remission is defined as MADRS ≤10. Response is defined as a reduction of >/=50% of MADRS baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Medhat M Bassiony, Professor, Principal Investigator — Zagazig University; Usama M Youssef, Professor, Study Director — Zagazig University; Ghada M Salah El-Deen, Professor, Study Director — Zagazig University; Hayam M El-Gohary, Professor, Study Director — Zagazig University; Alaa E Zayed, Ass.Lecturer, Study Director — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No